CLINICAL TRIAL: NCT04732793
Title: A Prospective, Active Controlled, Randomised, Parallel Group, Double Blind, Multicentre Study to Assess the Safety and Effectiveness of Hyruan ONE Versus a Comparator for the Treatment of Knee Osteoarthritis in Europe
Brief Title: To Assess the Safety and Effectiveness of Hyruan ONE Versus a Comparator for the Treatment of Knee Osteoarthritis in Europe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-HACL026
Record Dates: First submitted 2021-01-07; First posted 2021-02-01 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis (OA) of the Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyruan ONE® (Experimental)
  Interventions: Device: Hyruan ONE®
- Durolane® (Active Comparator)
  Interventions: Device: Durolane®

INTERVENTIONS:
Device: Hyruan ONE® — For use as a symptomatic treatment of osteoarthritis (OA) of the knee
  Arms: Hyruan ONE®
Device: Durolane® — For use as a symptomatic treatment of osteoarthritis (OA) of the knee
  Arms: Durolane®

SUMMARY:
To Assess the Safety and Effectiveness of Hyruan ONE versus a Comparator for the Treatment of Knee Osteoarthritis in Europe

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥40 years old.
2. Subject has radiographic evidence of mild-to-moderate OA (Kellgren Lawrence Scale grade II III) in one or both knees. Radiographs to be taken within 12 months prior to the Screening visit.
3. Subject has OA pain in the target knee despite conservative physical treatments and/or analgesics.

Exclusion Criteria:

1. Subject has rheumatoid arthritis or other inflammatory metabolic arthritis.
2. Subject has a documented history of hypersensitivity to HA.
3. Subject has a documented infection or severe inflammation of the target knee joint.
4. Subject has a skin disease in the area of the injection site.
5. Subject has a clinically apparently tense effusion of the target knee on examination determined by either a positive bulge sign or positive ballottement of the patella (patellar tap).
6. Subject has chronic pain requiring chronic ongoing analgesic therapy that confounds the measurement of pain in the target knee.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
The change in the WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index) Likert pain subscore | from Baseline to 13 weeks post injection.
  The WOMAC Likert Index measures 3 separate dimensions: pain, stiffness, and function. The subject will self assess the level of pain in the target knee joint for the prior 48 hours (5 questions), the level of difficulty of performing daily activities (17 questions), and the level of stiffness (2 questions) using the WOMAC Likert Questionnaire (24 total questions; 4 points/question).
  Each item of the WOMAC Likert Index will be assessed using the scale of 0=none, 1=a little, 2=moderate, 3=severe, 4=very severe. The aggregate total score that can result for each scale is as follows:
  Pain = 0-20 Stiffness = 0-8 Physical function = 0-68.

CONTACTS AND LOCATIONS:
Locations (1):
- Lubelskie Centrum Diagnostyczne, Świdnik, Poland